CLINICAL TRIAL: NCT04532528
Title: Relationship of Advanced Holding Education and ADherence on Antithrombotic in Younger SPAF Patients
Brief Title: ReAHEAD: A Study to Find Out Whether Education Improves Adherence to Dabigatran in People With Atrial Fibrillation Who Are Younger Than 75 Years
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0304
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard of care (SOC) only: This group includes Atrial Fibrillation (AF) patients diagnosed within 1 month, under 75 years old, and newly prescribed dabigatran on physician's decision based on local labelling.
  Interventions: Drug: Dabigatran
- SOC with advanced educational intervention: This group includes Atrial Fibrillation (AF) patients diagnosed within 1 month, under 75 years old, and newly prescribed dabigatran on physician's decision based on local labelling who also received advance educational intervention.
  The educational intervention was based on material of the "Shared decision making of treatment of New Oral AntiCoagulants (NOAC) in AF patients" and "Atrial Fibrillation Patient Care in Hospitals". The educational materials were delivered after baseline and at their 3, 6, 9, and 12 months visit.
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran — Dabigatran

SUMMARY:
Lifelong oral anticoagulant (OAC) therapy is the preferred treatment for the prevention of thromboembolic events in the majority of patients with Atrial Fibrillation (AF). Adherence to medication is essential for valid treatment for OAC therapy.

The study aims to explore whether the advanced educational intervention would improve the adherence to dabigatran.

ELIGIBILITY:
Inclusion Criteria:

Patients can be included if ALL the following criteria are met:

1. Provide written informed consent prior to participation
2. Female or male adult patients aged ≥ 20 years and < 75 years, newly diagnosed with non-valvular atrial fibrillation (NVAF) within 1 month and has newly prescribed with dabigatran on physician's decision before study enrolment.

Exclusion Criteria:

Patients should not be included if ANY ONE of the following criteria is met:

1. Contraindication to the use of dabigatran (i.e., active pathological bleeding, history of a serious hypersensitivity reaction to dabigatran [e.g., anaphylactic reaction or anaphylactic shock], severely impaired renal function [Creatinine clearance rate (Ccr) < 30 mL/min], hemorrhagic manifestations, bleeding diathesis, mechanical prosthetic heart valve, congenital or acquired coagulation disorders, organic lesions with bleeding tendency, or concomitantly use systemic ketoconazole, cyclosporine, and itraconazole)
2. Participate in other interventional trials currently or in the past 30 days

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients newly diagnosed with AF within 1 month, under 75 years old, and newly prescribed with dabigatran on physician's decision per local labelling will be equally randomized to receive standard of care (routine clinical practice) or standard of care (routine clinical practice) with advanced educational intervention.
Sampling Method: Probability Sample
Enrollment: 897 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- Taiwan (23):
  - Chia-Yi Christian Hospital, Chia-Yi City
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi City
  - National Taiwan University Hospital-Hsin-Chu Branch, Hsinchu
  - Buddhist Tzu Chi General Hospital, Hualien City
  - Kaohsiung Municipal Da-Tung Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - Pingtung Christian Hospital, Pingtung City
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - Kuang-Tien General Hospital, Taichung
  - NCKUH, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital(Linkou), Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Chu CS, Tsai CT, Huang CY, Li CH, Tsai HL, Liu YB, Liu JC, Chang HR, Lin WS, Chao TF, Tsao TP, Shih JY, Chong JT, Huang SC, Wu CC, Lin CS, Shih CC, Cheng CI, Chao TH, Chiang CH, Huang CH, Chien CY, Lei WY, Lin KR, Chu PH, Lin TH. The RElationship of Advanced Education and ADherence (ReAHEAD) on antithrombotic in younger patients with non-valvular atrial fibrillation in Taiwan. J Formos Med Assoc. 2025 Oct 13:S0929-6646(25)00529-7. doi: 10.1016/j.jfma.2025.10.002. Online ahead of print. PMID 41087222
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A retrospective cohort data analysis was conducted to assess the impact of an advanced educational intervention on the adherence to dabigatran in newly diagnosed atrial fibrillation adult patients under 75 years old in Taiwan.
Pre-assignment Details: Only participants that met all inclusion and none of the exclusion criteria were included. Participants were equally randomized in two cohorts: 'standard of care' and 'standard of care with advanced educational intervention'. Out of the 897 screened participants only 873 met the eligibility criteria and were included in the study.
Groups:
- SOC With Advanced Educational Intervention: This group includes Atrial Fibrillation (AF) patients diagnosed within 1 month, under 75 years old, and newly prescribed dabigatran on physician's decision based on local labelling who also received advance educational intervention.
  The educational intervention was based on material of the "Shared decision making of treatment of New Oral Anti Coagulants (NOAC) in AF patients" and "Atrial Fibrillation Patient Care in Hospitals". The educational materials were delivered after baseline and at their 3, 6, 9, and 12 months visit.
Period: Overall Study
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Started (Subjects who started the study.) | 441 | 432
3 Months (Subjects who completed the 3 months visit.) | 368 | 366
6 Months (Subjects who completed the 6 months visit.) | 308 | 312
9 Months (Subjects who completed the 9 months visit.) | 286 | 266
12 Months (Subjects who completed the 12 months visit.) | 271 | 246
Completed (Subjects who completed the study completion visit.) | 269 | 243
Not Completed | 172 | 189
Not completed — Adverse Event | 12 | 17
Not completed — Withdrawal of consent | 16 | 17
Not completed — Participant stop Dabigatran during the 12-month study period | 22 | 24
Not completed — Lost to Follow-up | 69 | 68
Not completed — Administrative problems | 12 | 14
Not completed — Death | 3 | 3
Not completed — Other | 38 | 46

BASELINE CHARACTERISTICS:
Population: Cohort of newly diagnosed Atrial Fibrillation (AF) adult patients who were under 75 years old and were prescribed dabigatran.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention | Total
Number analyzed (Participants) | 441 | 432 | 873
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (7.70) | 64.7 (7.49) | 65.0 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 167 | 348
  Male | 260 | 265 | 525
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Taiwanese | 441 | 430 | 871
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With High (MMAS-8 Score: 8 Points) Adherence to Dabigatran Treatment at Month 12 in Patients With and Without Advanced Educational Intervention
Description: Number of patients with high adherence to dabigatran treatment at month 12 in patients with and without advanced educational intervention was assessed by the Morisky 8-Item Medication Adherence Questionnaire (MMAS-8). A high adherence was defined as achieving a MMAS-8 score of 8 Points.
  The MMAS-8 is an 8-item structured, self-report measure that assesses medication adherence. The total score ranges from 0 to 8 with a higher score indicating a higher adherence.
  The validated Chinese MMAS-8 was used to evaluate the adherence to dabigatran at baseline and every follow-up visit. Patients were considered to have low adherence with scores of 0 to 5, medium adherence with scores of 6 to 7, and high adherence with a score of 8.
Time Frame: at 12 months
Population: Newly diagnosed Atrial Fibrillation (AF) patients who received dabigatran with and without advanced educational intervention who had high adherence to dabigatran. Arms were mutually exclusive. Only patients with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 271 | 246
Participants | 199 | 181
Statistical Analysis 1: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; Test type: Other — No formal hypotheses were tested; p = 0.9701, Chi-squared

2. Secondary Outcome: Number of Patients With High (MMAS-8 Score: 8 Points) Adherence to Dabigatran Treatment at 3, 6, and 9 Months in Patients With and Without Advanced Educational Intervention
Description: Number of patients with high adherence to dabigatran treatment at 3, 6, and 9 months in patients with and without advanced educational intervention was assessed by the Morisky 8-Item Medication Adherence Questionnaire (MMAS-8). A high adherence was defined as achieving a MMAS-8 score of 8 Points.
  The MMAS-8 is an 8-item structured, self-report measure that assesses medication adherence. The total score ranges from 0 to 8 with a higher score indicating a higher adherence.
  The validated Chinese MMAS-8 was used to evaluate the adherence to dabigatran at baseline and every follow-up visit. Patients were considered to have low adherence with scores of 0 to 5, medium adherence with scores of 6 to 7, and high adherence with a score of 8.
Time Frame: at 3, 6, and 9 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 363 | 364
Participants
  At 3 months | 224 | 229
  At 6 months: number analyzed (Participants) | 300 | 303
  At 6 months | 199 | 218
  At 9 months: number analyzed (Participants) | 284 | 262
  At 9 months | 204 | 184
Statistical Analysis 1: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 3 months only; Test type: Other — No formal hypotheses were tested; p = 0.7376, Chi-squared
Statistical Analysis 2: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 6 months only; Test type: Other — No formal hypotheses were tested; p = 0.1356, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 9 months only; Test type: Other — No formal hypotheses were tested; p = 0.6800, Chi-squared

3. Secondary Outcome: Number of Patients With Medium (MMAS-8 Score: 6 to 7 Points) Adherence to Dabigatran Treatment at 3, 6, 9, and 12 Months in Patients With and Without Advanced Educational Intervention
Description: Number of patients with medium adherence to dabigatran treatment at 3, 6, 9, and 12 months in patients with and without advanced educational intervention was assessed by the Morisky 8-Item Medication Adherence Questionnaire (MMAS-8). A medium adherence was defined as achieving a MMAS-8 score of 6 or 7 points.
  The MMAS-8 is an 8-item structured, self-report measure that assesses medication adherence. The total score ranges from 0 to 8 with a higher score indicating a higher adherence.
  The validated Chinese MMAS-8 was used to evaluate the adherence to dabigatran at baseline and every follow-up visit. Patients were considered to have low adherence with scores of 0 to 5, medium adherence with scores of 6 to 7, and high adherence with a score of 8.
Time Frame: At 3, 6, 9, and 12 months
Population: Newly diagnosed Atrial Fibrillation (AF) patients who received dabigatran with and without advanced educational intervention who had medium adherence to dabigatran. Arms were mutually exclusive. Only patients with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 363 | 364
Participants
  At 3 months | 83 | 77
  At 6 months: number analyzed (Participants) | 300 | 303
  At 6 months | 66 | 57
  At 9 months: number analyzed (Participants) | 284 | 262
  At 9 months | 52 | 53
  At 12 months: number analyzed (Participants) | 271 | 246
  At 12 months | 50 | 51
Statistical Analysis 1: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 3 months only; Test type: Other — No formal hypotheses were tested; p = 0.5777, Chi-squared
Statistical Analysis 2: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 6 months only; Test type: Other — No formal hypotheses were tested; p = 0.3313, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 9 months only; Test type: Other — No formal hypotheses was tested; p = 0.5697, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 12 months only; Test type: Other — No formal hypotheses were tested; p = 0.5135, Chi-squared

4. Secondary Outcome: Number of Patients With Low (MMAS-8 Score: 0 to 5 Points) Adherence to Dabigatran Treatment at 3, 6, 9, and 12 Months in Patients With and Without Advanced Educational Intervention
Description: Number of patients with low adherence to dabigatran treatment at 3, 6, 9, and 12 months in patients with and without advanced educational intervention was assessed by the Morisky 8-Item Medication Adherence Questionnaire (MMAS-8). A low adherence was defined as achieving a MMAS-8 score of 0, 1, 2, 3, 4, or 5 points.
  The MMAS-8 is an 8-item structured, self-report measure that assesses medication adherence. The total score ranges from 0 to 8 with a higher score indicating a higher adherence.
  The validated Chinese MMAS-8 was used to evaluate the adherence to dabigatran at baseline and every follow-up visit. Patients were considered to have low adherence with scores of 0 to 5, medium adherence with scores of 6 to 7, and high adherence with a score of 8.
Time Frame: At 3, 6, 9, and 12 months
Population: Newly diagnosed Atrial Fibrillation (AF) patients who received dabigatran with and without advanced educational intervention who had low adherence to dabigatran. Arms were mutually exclusive. Only patients with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 363 | 364
Participants
  At 3 months | 56 | 58
  At 6 months: number analyzed (Participants) | 300 | 303
  At 6 months | 35 | 28
  At 9 months: number analyzed (Participants) | 284 | 262
  At 9 months | 28 | 25
  At 12 months: number analyzed (Participants) | 271 | 246
  At 12 months | 22 | 14
Statistical Analysis 1: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 3 months only; Test type: Other — No formal hypotheses were tested; p = 0.8509, Chi-squared
Statistical Analysis 2: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 6 months only; Test type: Other — No formal hypotheses were tested; p = 0.3302, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 9 months only; Test type: Other — No formal hypotheses was tested; p = 0.9005, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 12 months only; Test type: Other — No formal hypotheses were tested; p = 0.2789, Chi-squared

5. Secondary Outcome: Mean MMAS-8 Score at 3, 6, 9, and 12 Months in Patients With and Without Advanced Educational Intervention
Description: Mean Morisky 8-Item Medication Adherence Questionnaire (MMAS-8) score at 3, 6, 9, and 12 months in patients with and without advanced educational intervention.
  The MMAS-8 is an 8-item structured, self-report measure that assesses medication adherence. The total score ranges from 0 to 8 with a higher score indicating a higher adherence.
  The validated Chinese MMAS-8 was used to evaluate the adherence to dabigatran at baseline and every follow-up visit. Patients were considered to have low adherence with scores of 0 to 5, medium adherence with scores of 6 to 7, and high adherence with a score of 8.
Time Frame: At 3, 6, 9, and 12 months
Population: Newly diagnosed Atrial Fibrillation (AF) patients who received dabigatran with and without advanced educational intervention. Arms were mutually exclusive. Only patients with available data were included in this analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 363 | 364
Score on a scale
  At 3 months | 7.0 (1.65) | 7.0 (1.72)
  At 6 months: number analyzed (Participants) | 300 | 303
  At 6 months | 7.2 (1.41) | 7.3 (1.38)
  At 9 months: number analyzed (Participants) | 284 | 262
  At 9 months | 7.4 (1.25) | 7.3 (1.27)
  At 12 months: number analyzed (Participants) | 271 | 246
  At 12 months | 7.4 (1.21) | 7.5 (1.07)
Statistical Analysis 1: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 3 months only; Test type: Other — No formal hypotheses were tested; p = 0.6670, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 6 months only; Test type: Other; p = 0.1285, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 9 months only; Test type: Other — No formal hypotheses was tested; p = 0.7151, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Standard of Care (SOC) Only vs SOC With Advanced Educational Intervention; At 12 months only; Test type: Other — No formal hypotheses were tested; p = 0.8030, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Patients Who Discontinued Treatment With Dabigatran in Patients With and Without Advanced Educational Intervention
Description: Number of patients who discontinued treatment with dabigatran in patients with and without advanced educational intervention.
Time Frame: up to 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 440 | 431
Participants
  Yes | 167 | 181
  No | 225 | 213
  Not done | 48 | 37

7. Secondary Outcome: Number of Patients Who Discontinued Treatment With Dabigatran and Reasons Why They Discontinued in Patients With and Without Advanced Educational Intervention
Description: Number of patients who discontinued treatment with dabigatran and reasons why they discontinued in patients with and without advanced educational intervention.
Time Frame: up to 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 167 | 181
Participants
  Switched to other treatment | 60 | 70
  Other | 107 | 111

8. Secondary Outcome: Number of Patients Who Switched Treatment With Dabigatran and Reasons Why They Switched in Patients With and Without Advanced Educational Intervention
Description: Number of patients who switched treatment with dabigatran and reasons why they switched in patients with and without advanced educational intervention
Time Frame: up to 12 months
Population: Newly diagnosed Atrial Fibrillation (AF) patients who received dabigatran with and without advanced educational intervention and then switched treatment. Arms were mutually exclusive. Only patients with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
Number analyzed (Participants) | 60 | 70
Participants
  Adverse event | 12 | 13
  Inconvenience | 3 | 3
  Cost | 1 | 0
  Treatment failure | 4 | 8
  Other reasons | 40 | 46

ADVERSE EVENTS:
Time Frame: From baseline up to 12 months All cause mortality adverse events were collected also after the subjects withdrew from the study.
Description: Subject who withdraw or discontinue the study due to adverse events which caused death and were reported in safety reports were also counted in All-Cause Mortality-Total Number Affected.
Arm/Group | Standard of Care (SOC) Only | SOC With Advanced Educational Intervention
All-Cause Mortality (participants affected / at risk) | 3/441 | 5/432
Serious Adverse Events (participants affected / at risk) | 4/441 | 5/432
Other Adverse Events (participants affected / at risk) | 0/441 | 0/432
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (SOC) Only (N=441) | SOC With Advanced Educational Intervention (N=432)
Cardiac arrest (Cardiac disorders) | 0 | 1
Death (General disorders) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Natural killer-cell lymphoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Document date is not required in the title page of the protocol/SEAP according to Boehringer Ingelheim internal policy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04532528/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04532528/SAP_001.pdf